CLINICAL TRIAL: NCT05926362
Title: Capillary-Venous Paired Data Collection
Acronym: CaVeP-DC
Status: Not yet recruiting | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS: 329382
Record Dates: First submitted 2023-05-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Capillary-venous paired data collection.

DETAILED DESCRIPTION:
An iterative data collection study to continuously assess the performance of our Entia Liberty device with cancer patients. Our device enables a full blood count from a finger prick sample. The participants enrolled in the study will attend the study site for their routine venepuncture blood test. Once enrolled, they will have a finger prick test obtained by a Healthcare Professional (trained member of the clinical research team) to be tested on an Entia Liberty device. Within 4 hours of that same participant's routine venepuncture, a small amount of blood from the venepuncture will be also tested on a second Entia Liberty device in the laboratory. All the results from the capillary finger prick Liberty test, routine venepuncture blood test (gold standard reference method) and the venous blood Liberty test will be compared against each other to regularly assess that the improvements made on the measurement system of the device is sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old at the time of study entry
* Currently receiving standard of care systemic anti-cancer therapy (chemotherapy, immunotherapy, endocrine and targeted therapy) for solid organ malignancy and has received at least one cycle of treatment
* Scheduled to be undergoing routine venous laboratory blood tests as part of standard of care
* Can provide written informed consent

Exclusion Criteria:

* History of haematological malignancy
* Inadequate use and understanding of the English language, requiring a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are currently receiving standard of care systemic anti-cancer therapy (chemotherapy, immunotherapy, endocrine and targeted therapy) for solid organ malignancy and have received at least one cycle.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Coefficient of Variance of the difference between the lab results and the Liberty results | 3 years
  the coefficient of variance (CV) between the lab results and the liberty results would be compared. a lower CV value signifies a better performance of our device.

IPD SHARING:
Plan to Share IPD: No
It is not planned to make individual participant data (IPD) available to other researchers.